CLINICAL TRIAL: NCT02221518
Title: Control & Reward Circuits as Targets for Repetitive Thoughts and Behaviors
Brief Title: Control and Reward Circuits in Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Helen Blair Simpson, Professor of Psychiatry-Columbia University Medical Center, Columbia University; Director of Anxiety Disorders Clinic & Center for OCD and Related Disorders, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: #7000/R01MH104648-01
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with OCD (Experimental): Behavioral: Exposure & Response Prevention (EX/RP)
  Interventions: Behavioral: Exposure & Response Prevention (EX/RP)

INTERVENTIONS:
Behavioral: Exposure & Response Prevention (EX/RP) — Exposure and Response Prevention (EX/RP) is a type of Cognitive Behavioral Treatment for treating OCD.

SUMMARY:
The purpose of this study is to examine the brain functioning of OCD patients and healthy controls before and after treatment with Exposure and Response Prevention (EXRP) therapy.

DETAILED DESCRIPTION:
The capacity to coordinate thoughts and actions to execute goal-directed behaviors (cognitive control) and the capacity to anticipate, respond to, and learn from reward (reward processing) are key processes for human behavior. Dysfunction in these processes has been hypothesized to contribute to repetitive thoughts and behaviors in many disorders, including obsessive-compulsive disorder (OCD), Tourette Syndrome (TS), and eating disorders. We will use multimodal imaging to investigate neural circuits that support cognitive control and reward processing, using OCD as a model system. The short-term goal is to clarify how circuit-based abnormalities contribute to repetitive thoughts/behaviors; these data will inform future transdiagnostic studies. The long-term goal is to identify control and reward circuit-abnormalities as targets for new transdiagnostic treatments.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Male and females with OCD aged 18-55
* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Diagnosis of OCD
* Not on psychotropic medication

Exclusion Criteria for Patients:

* Presence of metallic devices or dental braces in the body that are contraindicators for MR imaging
* Comorbid psychiatric conditions that significantly elevate the risk of study participation (e.g. psychotic disorders, bipolar disorder, evidence of dementia or other cognitive disorder, suicidality)
* Unstable medical conditions that need attention and would make participation in the study unsafe (e.g. very high blood pressure)
* Use of psychotropic medication
* Females who are pregnant or post-menopausal

Inclusion Criteria for Healthy Volunteers

- Male and females aged 18-55

Exclusion Criteria for Healthy Volunteers

* Presence of metallic devices or dental braces in the body that are contraindicators for MR imaging
* Any psychiatric diagnosis
* Use of psychotropic medication
* Diagnosis of OCD in a first degree relative
* Females who are pregnant or post-menopausal
* Unstable medical conditions that need attention and would make participation in the study unsafe (e.g. very high blood pressure)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in brain activation (fMRI) and fractional anisotropy (Diffusion tensor imaging) after therapy | Baseline & approximately 10 weeks later

SECONDARY OUTCOMES:
Change in reaction times and correct responses on Stop signal reaction time task | Baseline and approximately 10 weeks later, at second scan

CONTACTS AND LOCATIONS:
Overall Officials: Blair Simpson, MD, Ph.D, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- NY State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Wheaton MG, Kalanthroff E, Mandel M, Marsh R, Simpson HB. Neurocognitive performance in obsessive-compulsive disorder before and after treatment with cognitive behavioral therapy. J Behav Ther Exp Psychiatry. 2025 Jun;87:102019. doi: 10.1016/j.jbtep.2025.102019. Epub 2025 Jan 20. PMID 39879875
- [Derived] Shi TC, Pagliaccio D, Cyr M, Simpson HB, Marsh R. Network-based functional connectivity predicts response to exposure therapy in unmedicated adults with obsessive-compulsive disorder. Neuropsychopharmacology. 2021 Apr;46(5):1035-1044. doi: 10.1038/s41386-020-00929-9. Epub 2021 Jan 14. PMID 33446895
- [Derived] Pagliaccio D, Middleton R, Hezel D, Steinman S, Snorrason I, Gershkovich M, Campeas R, Pinto A, Van Meter P, Simpson HB, Marsh R. Task-based fMRI predicts response and remission to exposure therapy in obsessive-compulsive disorder. Proc Natl Acad Sci U S A. 2019 Oct 8;116(41):20346-20353. doi: 10.1073/pnas.1909199116. Epub 2019 Sep 23. PMID 31548396